CLINICAL TRIAL: NCT03108313
Title: Role of Aloe Vera Versus Fluoride Toothpaste in Changing High to Low Salivary Bacterial Count :Randomized Controlled Trial
Brief Title: Role of Aloe Vera Versus Fluoride Toothpaste in Changing High to Low Salivary Bacterial Count
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Neven Ahmed Ebrahim, principal investigator, resident at conservative department, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CEBC-CU-2017-30-16
Record Dates: First submitted 2017-03-29; First posted 2017-04-11 (Actual); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Caries, Dental
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: A participant will generate the random allocation sequence. The researcher will enroll the patients but an unbiased participant will assign the intervention/Control identification procedures .The participants will be blinded to intervention/control assessment methods. Also, it will not be allowed among the examiners to exchange any information throughout the entire study period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- aloe vera toothpaste (Experimental): aloe vera toothpaste isa will be administrated 2 times per day for 30 days and salivary bacterial count will be tested before the use of toothpaste the after 15 days and 30 days
  Interventions: Drug: aloe vera toothpaste
- fluoride toothpaste (Active Comparator): fluoride toothpaste isa herbal toothpaste will be administrated 2 times per day for 30 days and salivary bacterial count will be tested before the use of toothpaste the after 15 days and 30 days
  Interventions: Drug: fluoride toothpaste

INTERVENTIONS:
Drug: aloe vera toothpaste — herbal toothpaste used to decrease salivary streptococcus bacterial count
  Other Names: aloe dent toothpaste; aloe dent
  Arms: aloe vera toothpaste
Drug: fluoride toothpaste — chemical toothpaste used to decrease salivary streptococcus bacterial count
  Other Names: signal toothpaste
  Arms: fluoride toothpaste

SUMMARY:
Patient's salivary bacterial count will be evaluated , then the patient will bbe instructed to follow oral hygiene measures including the use of aloe vera toothpaste or fluoride toothpaste , the after 15 days and 30 days the patient's salivary bacterial count will be evaluated another time.

DETAILED DESCRIPTION:
Variables of study:

Each patient will be instructed to follow oral hygiene measures including aloe vera or fluoride toothpaste

Outcomes:

Salivary bacterial count will be evaluated using Mitis salivarius agar plates before the use of the aloe vera toothpaste then after 15 days then after 30 days .

Participant timeline:

Enrolment Baseline assessment 15 days 30 days

(1st visit ) (2nd visit) (3rd visit )

II.6.Sample size calculation :

Based on previous study , the mean percent change reduction in bacterial count was 3+4 . using power 80 % and 5 % significance level , we will need to study 29 in each group to be able to reject the null hypothesis that the population means of the experimental and control groups are equal with probability (power) 0.8. The Type I probability associated with this test of this null hypothesis is 0.05.

Recruitment & Recruitment Strategy:

Screening of patients that come to the conservative dentistry department seeking dental care will continue until the target population is achieved. The patients will be subjected to full examination and diagnosis using dental charts. Once the patients that are potentially eligible for this study are identified, they will be contacted by the research investigator who will explain the study and ascertains the patient's interest. Randomization and assignment of interventions:

Randomization will be done according to a check list including the number of participants divided into 2 groups according to interventions/Control assessment method

Allocation sequence generation:

The allocation sequence will be generated using (www.randomization.com).

Allocation concealment mechanism:

A checklist will be designed to identify each assessment method.

Implementation A participant will generate the random allocation sequence. The researcher will enroll the patients but an unbiased participant will assign the intervention/Control identification procedures to respective teeth.

Blinding:

The participants will be blinded to intervention/control assessment methods. Also, it will not be allowed amongst the examiners to exchange any information throughout the entire study period.

Data collection methods:

High caries index will be assessed 3 times , at base line , then 15 days and 30 days.

Funding:

The research will be self-funded by the researcher.

ELIGIBILITY:
Inclusion Criteria:

* Patients should have poor oral hygiene.
* Patients should have high bacterial count

Exclusion Criteria:

* Patients with a compromised medical history.
* Severe or active periodontal disease .

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2017-03-03 (Actual); Primary Completion 2018-04-30 (Estimated); Study Completion 2018-04-30 (Estimated)

PRIMARY OUTCOMES:
salivary bacterial count | average of 30 days
  will be done using mitis salivarius agar plate

CONTACTS AND LOCATIONS:
Overall Officials: Amira Farid, PHD, Study Director — professor at conservative department cairo university; Rasha Rafaat, PHD, Study Chair — lecturer at conservative department cairo university
Locations (1):
- Neven Ahmed Ebrahim, Cairo, Heliopolis, Egypt

IPD SHARING:
Plan to Share IPD: Yes
publishing the data at egyptian dental journal

REFERENCES:
- [Background] Bhati N, Jaidka S, Somani R. Evaluation of antimicrobial efficacy of Aloe vera and Meswak containing dentifrices with fluoridated dentifrice: An in vivo study. J Int Soc Prev Community Dent. 2015 Sep-Oct;5(5):394-9. doi: 10.4103/2231-0762.165924. PMID 26539392